CLINICAL TRIAL: NCT03250624
Title: Safety and Efficacy of CD5024 0.3% Cream in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RD.03.SPR.109696
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD5024 0.3% cream (Experimental)
  Interventions: Drug: CD5024 0.3% cream
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD5024 0.3% cream — Participants applied CD5024 0.3% cream topically in the evening to the affected areas as a thin film corresponding to approximately 2 milligrams per centimeter square (mg/cm^2) once daily for 6 weeks.
  Other Names: Ivermectin
  Arms: CD5024 0.3% cream
Drug: Placebo — Participants applied placebo matched to CD5024 0.3% cream topically in the evening to the affected areas as a thin film corresponding to approximately 2 mg/cm^2 once daily for 6 weeks.
  Arms: Placebo

SUMMARY:
Exploratory, multi-centric, randomized, vehicle-controlled, investigator-blind, parallel group study, involved participants with chronic lesions of Atopic Dermatitis (AD) to evaluate the local and systemic safety of CD5024 0.3% cream over a 6-week treatment period compared to its vehicle.

DETAILED DESCRIPTION:
Study application was performed once daily, 7 days a week for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The participant was a male or female aged 18 to 60 years old inclusive at Screening.
2. The participant presented with a total body surface area (tBSA) less than or equal to (>=) 2 square meter (m^2) at Screening.
3. The participant had atopic dermatitis for at least 6 months prior to Day 1. The clinical diagnosis of atopic dermatitis must be confirmed with the criteria of Hanifin and Rajka at the screening visit.
4. Atopic dermatitis must be stable for at least one month before the screening visit (according to participant).
5. The participant had a Body Surface Area (BSA) affected by AD ranging from 1% inclusive to 10% inclusive at Day 1, excluding scalp and genitals.
6. The participant had an overall Investigator's Global Assessment (IGA) score of 3 (moderate) at Day 1;

Exclusion Criteria:

1. The participant was a pregnant female, is breastfeeding or intends to conceive a child during the study,
2. The participant had any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with the interpretation of the clinical trial results (e.g. extensive scaring or pigmented lesion in a treated area), and/or put the participant at significant risk according to Investigator's judgment if he/she participates in the clinical trial (e.g. active cancer, AIDS, insulin-dependent diabetes…) at Screening or Day 1.
3. The participant presented with an acute flare of AD at Day 1.
4. The participant had active cutaneous bacterial or viral infection in any treated area at baseline (e.g. clinically infected AD) at Screening or Day 1.
5. The participant had a history of confounding skin condition (e.g. psoriasis, erythroderma) or a history of Netherton syndrome at Screening.
6. The participant had a past history of serious persistent neurological disorders such as seizures, multiple sclerosis, or neurological signs or symptoms at Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Galderma Investigational Site (#8581), Mississauga, Ontario
  - Galderma Investigational Site (# 8338), Richmond Hill, Ontario
  - Galderma Investigational Site (#8587), Richmond Hill, Ontario
  - Galderma Investigational Site (# 8060), Windsor, Ontario
  - Galderma Investigational Site (#8089), Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 centers in Canada between 01 November 2016 and 26 June 2017.
Pre-assignment Details: A total of 101 participants were screened in the study. Out of which, 63 participants were randomized in a ratio of 1:1 to receive CD5024 0.3 percent (%) cream or its vehicle. Screen failures were mainly due to exclusion criteria met.
Groups:
- CD5024 0.3% Cream: Participants applied CD5024 0.3% cream topically in the evening to the affected areas as a thin film corresponding to approximately 2 milligrams per centimeters square (mg/cm^2) once daily for 6 weeks.
Period: Overall Study
Arm/Group | CD5024 0.3% Cream | Placebo
Started | 32 | 31
Completed | 30 | 24
Not Completed | 2 | 7
Not completed — Lack of Efficacy | 1 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) efficacy analysis set was defined as any participants who are randomized.
Groups:
- CD5024 0.3% Cream: Participants applied CD5024 0.3% cream topically in the evening to the affected areas as a thin film corresponding to approximately 2 mg/cm^2 once daily for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | CD5024 0.3% Cream | Placebo | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (9.19) | 30.0 (10.77) | 28.6 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 25 | 23 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicated the worse severity of AD.
  score on a scale | 5.341 (2.432) | 5.371 (2.652) | 5.356 (2.542)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score at Day 43
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum), with the higher scores indicated the worse severity of AD. All missing values were imputed by Last Observation Carried Forward (LOCF).
Time Frame: Baseline, Day 43
Population: The Intent-to-treat (ITT) efficacy analysis set was defined as any participant who were randomized.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 32 | 31
score on a scale | -2.64 (0.41) | -2.36 (0.44)
Statistical Analysis 1: Comparison: CD5024 0.3% Cream vs Placebo; Test type: Superiority; p = 0.632, ANCOVA; Least Square (LS) Mean Difference = -0.28, 95% CI 2-sided [-1.46 to 0.89]

2. Secondary Outcome: Percent Change From Baseline in EASI at Each Visit
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, induration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores indicated the worse severity of AD. All missing values were imputed by LOCF.
Time Frame: Baseline, Days 8,15, 22, 29, 36 and 43
Population: The ITT efficacy analysis set was defined as any participant who were randomized.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 32 | 31
percent change
  Day 8 | -8.7 (19.1) | -5.5 (39.6)
  Day 15 | -21.0 (37.5) | -10.7 (43.7)
  Day 22 | -29.1 (40.7) | -26.7 (35.8)
  Day 29 | -34.5 (59.9) | -21.0 (41.7)
  Day 36 | -43.1 (35.3) | -28.8 (44.7)
  Day 43 | -46.4 (38.8) | -24.6 (62.7)

3. Secondary Outcome: Percentage of Participants Who Achieved an Investigator Global Assessment (IGA) Score of 1 (Almost Clear) or 0 (Clear)
Description: IGA scale consisted of 5 grades (0-4) among which 0 = Clear (Minor, residual discoloration, no erythema or induration/papulation, no oozing/crusting), 1 = Almost clear (Trace, faint pink erythema with almost no induration/papulation and no oozing/crusting), 2 = Mild (Faint pink erythema with mild induration/papulation and no oozing/crusting), 3 = Moderate (Pink-red erythema with moderate induration/papulation and there may be some oozing/crusting.), 4 = Severe (Deep/bright red erythema with severe induration/papulation with oozing/crusting). Success rate was defined as percentage of participants who achieved an IGA score of 1 (almost clear) or 0 (Clear) at specified visits. All missing values were imputed by LOCF.
Time Frame: Days 8, 15, 22, 29, 36 and 43
Population: The ITT efficacy analysis set was defined as any participant who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 32 | 31
percentage of participants
  Day 8 | 0 | 3.23
  Day 15 | 3.13 | 6.45
  Day 22 | 9.38 | 9.68
  Day 29 | 15.6 | 6.45
  Day 36 | 21.9 | 16.1
  Day 43 | 37.5 | 9.68

4. Secondary Outcome: Percent Change From Baseline in Total Sum Score (TSS) at Each Visit
Description: The TSS was the sum of individual clinical severity scores for 5 signs of AD (erythema, induration/papulation, oozing/crusting, excoriation and lichenification). The severity of each sign was evaluated by using a 4-graded scale (0: none; 1: mild; 2: moderate; 3: severe). The total score ranges from 0 to 15, where higher score indicated worse severity of AD. All missing values were imputed by LOCF.
Time Frame: Baseline, Days 8, 15, 22, 29, 36 and 43
Population: The ITT efficacy analysis set was defined as any participant who were randomized.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 32 | 31
percent change
  Day 8 | -15.35 (4.51) | -17.30 (4.75)
  Day 15 | -27.94 (5.76) | -20.82 (6.07)
  Day 22 | -29.38 (6.23) | -33.57 (6.57)
  Day 29 | -37.23 (6.64) | -34.44 (6.99)
  Day 36 | -45.01 (6.75) | 42.24 (7.11)
  Day 43 | -47.63 (7.30) | -45.00 (7.69)

5. Secondary Outcome: Percent Change From Baseline in Modified Objective Scoring Atopic Dermatitis (SCORAD) at Each Visit
Description: SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with visual analog scale (VAS) where 0 is no itching or no trouble sleeping and 10 is unbearable itching or a lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. Higher scores indicated worse outcome. All missing values were imputed by LOCF.
Time Frame: Baseline, Days 8, 15, 22, 29, 36 and 43
Population: The ITT efficacy analysis set was defined as any participant who were randomized.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 32 | 31
percent change
  Day 8 | -16.28 (4.29) | -16.00 (4.52)
  Day 15 | -30.76 (5.51) | -20.49 (5.81)
  Day 22 | -32.02 (5.84) | -30.73 (6.16)
  Day 29 | -39.14 (6.51) | -31.81 (6.86)
  Day 36 | -46.38 (6.67) | -40.10 (7.03)
  Day 43 | -48.92 (7.26) | -41.48 (7.65)

6. Secondary Outcome: Change From Baseline in Pruritus Numerical Rating Scale (NRS) at Each Visit
Description: Pruritus NRS was a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 = 'no itch' and 10 = 'worst itch imaginable', where higher score indicated very severe itch. All missing values were imputed by LOCF.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5 and 6
Population: The ITT efficacy analysis set was defined as any participant who were randomized. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 31 | 29
score on a scale
  Week 1 | -0.2 (1.1) | -0.2 (1.4)
  Week 2 | -0.6 (1.9) | -0.3 (1.7)
  Week 3 | -0.7 (2.1) | -0.4 (1.9)
  Week 4 | -1.0 (2.3) | -0.3 (2.1)
  Week 5 | -1.0 (2.2) | -0.5 (2.0)
  Week 6 | -1.3 (2.4) | -0.6 (2.1)

7. Secondary Outcome: Change From Baseline in Pruritus Verbal Rating Scale (VRS) Score at Day 43
Description: Participants were asked for a response that best described their pruritus intensity in last 24 hours, to rate their itch using a list of adjectives describing different levels of symptom intensity rated on a scale of 0 to 3 that is (i.e.) 0 = No itch, 1 = low, 2 = Moderate and 3 = Severe, where higher score indicated very severe itch. All missing values were imputed by LOCF.
Time Frame: Baseline, Day 43
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CD5024 0.3% Cream | Placebo
Number analyzed (Participants) | 26 | 24
score on a scale | -.31 (0.79) | -.13 (0.74)

ADVERSE EVENTS:
Time Frame: Up to Week 9
Description: The Safety set included all randomized participants who applied/were administered the study drug(s) at least once.
Arm/Group | CD5024 0.3% Cream | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 16/32 | 21/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5024 0.3% Cream (N=32) | Placebo (N=31)
Nasopharyngitis (Infections and infestations) | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Folliculitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 2
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Eyelid pain (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03250624/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT03250624/SAP_001.pdf